CLINICAL TRIAL: NCT01187472
Title: Organ Preservation in the Multispeciality Therapy of Stage II-IV Locally Advanced Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 12145B
Record Dates: First submitted 2010-08-20; First posted 2010-08-24 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Head and Neck Cancer
Keywords: Head; neck; cancer; advanced; oral cavity; lip; larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms; Lymphoid Interstitial Pneumonia; Laryngeal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treated subjects: Subjects treated on a previous study of locally advanced head and neck cancer

SUMMARY:
This protocol was opened to collect long term survival information on subjects enrolled in a previous study which evaluated the impact of neoadjuvant chemotherapy and concomitant chemoradiotherapy with organ preserving optional surgery on overall survival, time to progression, pattern of disease recurrence in patient with locally advanced head and neck cancer. The last surviving subject was last treated in 1989, and was lost to follow up in 2010.

ELIGIBILITY:
Eligibility Criteria:

Eligibility Criteria:

Subjects previously enrolled in a treatment protocol for locally advanced head and neck cancer who met the following criteria:

1. Patients with Stage IV carcinoma of the nasal or oral cavity, nasopharynx pharynx, larynx, paranasal sinuses, cervical esophagus, or hypopharynx are eligible. Patients with Stage III carcinoma of the nasopharynx, base of tongue and hypopharynx are also eligible. Therapy is given with curative intent.

   Prior to entry in the study the resectability and standard treatment options for each patient will be determined during a joint evaluation by a team composed of an attending surgeon, a radiation oncologist and a medical oncologist. In addition the timing and feasibility of surgery will be determined in each patient prior to initiation of therapy. The unequivocal demonstration of distant metastasis confers in eligibility.
2. Measurable disease is not required, but all disease will be carefully evaluated.
3. Patients must have a histologically or cytologically confirmed diagnosis of squamous cell carcinoma, mucoepidermoid carcinoma or lymphoepithelioma.
4. Patients must have not received prior chemotherapy or radiotherapy.
5. Patients must have performance status of >60%
6. Patients must have a WBC count of >3.5, an ANC count >1500 and a platlet count of >100,000.
7. The serum creatinine must be equal to or less than 1.5 m/dlor the calculated creatinine clearance must exceed 50cc/min.
8. Patient must be free of significant infection or other severe complicating medical illness.
9. Pregnancy will constitute an absolute contraindication to entrance on this protocol.

Min Age: 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects enrolled on a previous head and neck cancer treatment protocol
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2003-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | Until Death
  To collect long term survival information on subjects treated on a previous protocol which evaluated the the impact of neoadjuvant chemotherapy and concomitant chemoradiotherapy with organ preserving optional surgery on overall survival, time to progression, and pattern of disease recurrence in patients with locally advanced head and neck cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Everett E Vokes, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States